CLINICAL TRIAL: NCT06125054
Title: Boosting and Guiding Neuroplasticity by Combining Ketamine with Neurofeedback-assisted Learning - Towards an Individualized and Integrated Pharmaco-psychotherapy for Cocaine Addiction
Brief Title: Ketamine and Neurofeedback-Training: Effects on Neuroplasticity in Cocaine Addiction
Acronym: Co-Boost
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. med. Marcus Herdener (Other)
Collaborators: University of Zurich (Other); University of Vienna (Other); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Marcus Herdener, Dr. med., Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Co-Boost_PUK_2022-01859
Record Dates: First submitted 2023-10-26; First posted 2023-11-09 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cocaine Use Disorder; Cocaine Dependence
Keywords: Cocaine; Cocaine Use; Ketamine; Reward Sensitivity; Glutamate; Placebo-controlled; Therapeutic effects; Mechanistic effects; Neurofeedback Training; realtime fMRI
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double blind, parallel group, single center study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- rt-fMRI NFT / Placebo (Experimental): Participants get real time neurofeedback based on an experimental regions' activity and receive a 0.9% saline solution (i.v.) over 40 minutes.
  Interventions: Drug: Placebo; Behavioral: real-time fMRI neurofeedback training
- rt-fMRI NFT / Ketamine (Experimental): Participants get real time neurofeedback based on an experimental regions' activity and receive 0.71mg ketamine (i.v.) per kilogram bodyweight.
  Interventions: Drug: Ketamine; Behavioral: real-time fMRI neurofeedback training
- sham NFT / Placebo (Placebo Comparator): Participants get a real time neurofeedback based on a control regions' activity, which serves as a sham region and receive a 0.9% saline solution (i.v.) over 40 minutes.
  Interventions: Drug: Placebo; Behavioral: sham real-time fMRI neurofeedback training
- sham NFT / Ketamine (Experimental): Participants get a real time neurofeedback based on a control regions' activity, which serves as a sham region and receive 0.71mg ketamine (i.v.) per kilogram bodyweight.
  Interventions: Drug: Ketamine; Behavioral: sham real-time fMRI neurofeedback training

INTERVENTIONS:
Drug: Ketamine — single dose of ketamine (0.71mg/kg bodyweight i.v. over 40 minutes)
  Arms: rt-fMRI NFT / Ketamine; sham NFT / Ketamine
Drug: Placebo — single dose of placebo (0.9% saline solution i.v. over 40 minutes)
  Other Names: 0.9% saline solution
  Arms: rt-fMRI NFT / Placebo; sham NFT / Placebo
Behavioral: real-time fMRI neurofeedback training — Real-time fMRI based neurofeedback over 20 minutes where participants are instructed to perform reward imagery. The feedback is based on an experimental region. The training is repeated three times.
  Arms: rt-fMRI NFT / Ketamine; rt-fMRI NFT / Placebo
Behavioral: sham real-time fMRI neurofeedback training — Sham real-time fMRI neurofeedback training over 20 minutes where participants are instructed to perform reward imagery. The feedback is based on a control region. The training is repeated three times.
  Arms: sham NFT / Ketamine; sham NFT / Placebo

SUMMARY:
The goal of this clinical trial is to learn about the effects of the combination of ketamine and realtime functional magnetic resonance imaging (fMRI) neurofeedback training in individuals with cocaine use disorder. The main questions the investigators aim to answer are:

* Can the investigators observe a positive, significant effect on percentage of cocaine use days of both interventions combined as well as stand alone interventions?
* Is there a significant transfer effect of the neurofeedback training?
* Is there a significant, ketamine-dependent change in glutamate levels in the nucleus accumbens?

Participants will be given ketamine and a realtime fMRI neurofeedback training. Both interventions are placebo-controlled. The investigators will compare the four intervention groups to investigate the effects of the stand-alone effects of the intervention and the combination of it.

DETAILED DESCRIPTION:
Cocaine is the most frequently used stimulant worldwide, and its consumption rate in Europe indicates a continuing upward trend. Cocaine use is associated with great harms for affected individuals, their families, and the society. Unfortunately, until today no pharmacotherapy has been approved for the treatment of cocaine use disorder (CUD) due to lack of efficacy of tested compounds.

The investigators therefore propose, to use latest advancements in proton magnetic resonance spectroscopy (1H-MRS) and real time functional magnetic resonance imaging neurofeedback training (rt-fMRI NFT) to develop a neurobiologically informed experimental approach for an individualized and integrated pharmaco-psychotherapy that has the potential to open new avenues for the treatment of CUD, and in addition, to be transferable to other neuropsychiatric conditions.

To improve the efficacy of psychotherapeutic interventions in individuals with CUD, the investigators recently developed an rt-fMRI NFT paradigm based on reward imagery to specifically modify maladaptive reward sensitivity by self-regulating the brain's reward circuits.

Furthermore, using a 1H-MRS technique, the investigators recently demonstrated that a disturbed glutamate homeostasis in the nucleus accumbens (NAcc), an important hub in the brain's reward system, characterizes cue-induced craving in CUD. This indicates that urgently needed novel pharmacotherapies for addiction treatment should target the glutamatergic system.

Thus, to restore the glutamate homeostasis and to boost learning effect of the reward imagery training, the investigators propose to combine reward imagery rt- fMRI NFT with the N-methyl-D-aspartate (NMDA) receptor antagonist ketamine, which has direct effects both on glutamatergic signaling and neuroplasticity and has shown therapeutic potential to reduce cocaine craving and cocaine us.

The investigators anticipate a) restoration of the glutamate homeostasis in the NAcc b) changes in maladaptive reward sensitivity resulting from rt-fMRI NFT and c) synergistic effects of the pharmacological and the psychotherapeutic effect due to the ketamine-induced neuroplasticity that might open a window of opportunity for imagery-based learning. The investigators hypothesize that these neurobiological adaptions induced by the described interventions underlie their therapeutic effects on cocaine craving and use.

The effects of ketamine and reward imagery rt-fMRI NFT in individuals with CUD will be tested in a randomized, placebo-controlled, double blind, parallel group study.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Male and female cocaine users 18 to 55 years of age
* diagnostic and statisical manual (DSM)-5 diagnosis of CUD
* Willingness to comply with the study protocol as explained by investigator
* Normal level of language comprehension (German or Swiss-German)

Exclusion Criteria:

* Current or lifetime psychotic disorders
* History of severe substance-induced psychosis
* Current or lifetime bipolar I or II disorders
* Current suicidality
* Previous suicide attempts during the last 2 years
* Current severe alcohol use disorder
* Current severe cannabis use disorder
* Current moderate or severe stimulant use disorder (other than cocaine)
* Current moderate or severe benzodiazepine use disorder
* Current opioid use disorder
* First-degree relatives with psychotic disorders
* Beck Depression Inventory Score greater than 25
* Unmedicated or unstable hypertension
* Severe illness (e. g. myocardial ischemia or arrythmias, severe pulmonary secretions, glaucoma, congestive heart failure or angina, significant renal or hepatic impairment)
* Acute infection (e. g. pulmonary or upper respiratory tract infection)
* Insufficient treated or uncorrected hyperthyroidism
* Severe central nervous system related traumas or disorders (e. g. stroke, cerebral trauma with loss of consciousness over more than 24h, epilepsy)
* Increased intracranial pressure
* Medication directly affecting glutamate signaling (e. g. anticonvulsant medication)
* Any unstable psychoactive medication (no changes in compounds within last 4 weeks before start of study)
* Pregnancy or lactation
* Women of childbearing potential with no use of medically accepted contraceptive (e. g.

condoms, contraceptive diaphragm, birth control pill, hormone injection, intrauterine device)

* BMI>35
* Allergy, hypersensitivity, or other adverse reaction to previous use of ketamine
* Contradictions to magnetic resonance imaging
* Concurrent participation in other clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Decrease in proportion of cocaine use days | Between 5 and 7 weeks after baseline (the first intervention visit)
  Between-group comparison of proportion of cocaine use days measured with Time-Line Follow-Back questionnaire for cocaine use on follow-up visit (t3).
Changes in fMRI signal of neurofeedback training | Between 1 and 2 weeks after baseline (the first neurofeedback training)
  Signal changes assessed with fMRI between the non-neurofeedback run 1 on Interention Visit I (t1) and run 3 on Intervention Visit II (t2).
Changes in accumbal glutamate levels | Before and during infusion (same day)
  Baseline and acute accumbal glutamate levels assessed with 1H-MRS on Intervention Visit I (t1).

SECONDARY OUTCOMES:
Changes in urine cocaine and cocaine metabolites | Baseline (screening visit) up to 19 weeks later (Follow-up Visit)
  Changes in cocaine and cocaine metabolites via urine analysis as objectified measure of cocaine use.
Cocaine craving | From baseline (screening visit) until 38 weeks later (Follow-up Survey)
  Changes in cocaine craving score assessed by the Obsessive Compulsive Cocaine Use Scale, ranging from 0 to 56, where higher scores indicate more problematic behavior and thoughts.
Severity of cocaine use disorder | From baseline (screening visit) until 38 weeks later (Follow-up Survey)
  Changes in severity of cocaine use disorder assessed by the Obsessive Compulsive Cocaine Use Scale, ranging from 0 to 56, where higher scores indicate more problematic behavior and thoughts.
Current motivation to change cocaine use behaviour | From baseline (screening visit) until 38 weeks later (Follow-up Survey)
  Changes in current motivation to change cocaine use behaviour assessed by an visual analogue scale ranging from 0 to 30 where higher scores indicate a higher motivation to change.
Hedonic capacity | From baseline (screening visit) until 38 weeks later (Follow-up Survey)
  Changes in hedonic capacity measured by the Trait Hedonic Capacity Scale, ranging from 16 to 80, where a higher score indicates a higher hedonic capacity.
Experience of pleasure across different domains | From baseline (screening visit) until 38 weeks later (Follow-up Survey)
  Changes in the experience of pleasure across different domains assessed by the Domains of Pleasure Scale, ranging from 0 to 210 where a higher score indicates a higher experience of pleasure.
Emotion regulation skills | Baseline (screening visit) and up to 19 weeks later (Follow-up Visit)
  Changes in emotion regulation skills measured with the Negative Mood Regulation expectancies Scale, ranging from 30 to 150 where higher scores indicate higher emotion regulation skills.
Depressive symptoms | Baseline (screening visit), up to 14 weeks later (Intervention Visit II), and up to 19 weeks later (Follow-up Visit)
  Changes in depressive symptoms measured with the Beck Depression Inventory. The scale ranges from 0 to 63 where higher scores indicate more severe depressive symptoms.
Perceived stress | Baseline (screening visit), up to 19 weeks later (Follow-up Visit), and up to 38 weeks later (Follow-up Survey)
  Changes in perceived stress assessed with a subscale of the Stress & Coping Inventory, ranging from 21 to 147 where higher scores indicate higher perceived stress.
Self-esteem | Baseline (screening visit), up to 14 weeks later (Intervention Visit II), up to 19 weeks later (Follow-up Visit), and up to 38 weeks later (Follow-up Survey)
  Changes in self-esteem assessed with the Rosenberg Self-esteem Scale, ranging from 0 to 30 where higher scores indicate a higher self-esteem.
Self-efficacy, optimism, and pessimism | Baseline (screening visit), up to 14 weeks later (Intervention Visit II), up to 19 weeks later (Follow-up Visit), and up to 38 weeks later (Follow-up Survey)
  Changes in Self-efficacy, optimism, and pessimism assessed with the Questionnaire for Self-efficacy, Optimism, and Pessimism (KSWOP-9), ranging from 9 to 36 where higher scores indicate higher self-efficacy, optimism, and pessimism, respectively.
Subjective effects of ketamine infusion | 2 hours post infusion
  Assess the acute subjective effects of the infusion with the Five-Dimension Altered State of Consciousness Questionnaire (5D-ASC), where the global score and each of the 11 subscales range from 0 to 100 and higher scores indicate the occurence of altered states of consciousness.
Effects of ketamine infusion on mystic experiences | 2 hours post infusion
  Assess the acute subjective effects of the infusion with the Hood's Mysticism Scale, ranging from 20 to 100 where higher scores indicate the occurence of mystic experiences.
Sustained changes in accumbal glutamate levels | Baseline (pre infusion, Intervention Visit I) and up to 2 weeks after infusion and neurofeedback training (Intervention Visit II)
  Assess sustained effects of the infusion and the neurofeedback training on baseline accumbal glutamate levels with 1H-MRS.
Glutamate levels during craving paradigm | Up to 2 weeks post infusion and neurofeedback training
  Assess the effects of the infusion and the neurofeedback training on glutamate levels measured by 1H-MRS during a craving paradigm.
Changes in Brain Derived Neurotrophic Factor | 0.5 hours pre infusion and 2 hours post infusion
  Assess changes in Brain Derived Neurotrophic Factor (BDNF) through blood analysis before and after the infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric University Hospital Zurich, University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Our data will be published on the website of Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the publication of our data.

REFERENCES:
- [Derived] Trippel AS, Gubser LP, Engeli EJE, Conradi J, Haugg A, Zoelch N, Herdener M. Co-Boost: boosting and guiding neuroplasticity by combining ketamine with neurofeedback-assisted learning-towards an individualised and integrated pharmaco-psychotherapy for cocaine addiction: study protocol for a randomised, placebo-controlled, double-blind, parallel-group, single-centre trial. Trials. 2025 Sep 25;26(1):354. doi: 10.1186/s13063-025-08982-9. PMID 40999531